CLINICAL TRIAL: NCT01685983
Title: A Phase 2 Open Label Study of Abiraterone Acetate (JNJ-212082) and Prednisolone in Patients With Advanced Prostate Cancer Who Have Failed Androgen Deprivation and Docetaxel-Based Chemotherapy.
Brief Title: A Study of Abiraterone Acetate (JNJ-212082) and Prednisolone in Patients With Advanced Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR100009; 212082PCR2007 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2012-09-12; First posted 2012-09-17 (Estimated); Results first posted 2016-05-23 (Estimated); Last update posted 2019-03-15 (Actual); Status verified 2019-02

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; Metastatic-castration resistant prostate cancer; Prostate specific antigen; Abiraterone acetate; JNJ-212082; Abiraterone; Prednisolone; Androgen Deprivation; Docetaxel-based chemotherapy
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Abiraterone Acetate; Prednisolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

ARMS (1):
- Abiraterone actetate and Prednisolone (Experimental)
  Interventions: Drug: Abiraterone acetate; Drug: Prednisolone

INTERVENTIONS:
Drug: Abiraterone acetate — Type=exact number, unit=mg, number=250, form=tablet, route=oral. Patients will receive 4 tablets of abiraterone acetate at least 1 hour before a meal or 2 hours after a meal any time up to 10 pm every day.
  Other Names: JNJ-212082
Drug: Prednisolone — Type=exact number, unit=mg, number=5, form=tablet, route=oral. Patients will receive 1 tablet of prednisolone twice daily.

SUMMARY:
The purpose of this study is to assess the safety and efficacy in Korea or Taiwan of oral abiraterone acetate and oral prednisolone in men with metastatic-castration resistant prostate cancer (mCRPC) and with disease progression following treatment with a docetaxel-containing chemotherapy.

DETAILED DESCRIPTION:
This is an open-label (all people know the identity of the intervention), multicenter, single arm (only one treatment group) study to evaluate the efficacy and safety of abiraterone acetate in patients with mCRPC. The study will be divided into screening phase (up to 28 days before enrollment), treatment phase including treatment cycles (each cycle of treatment will be 28 days), and follow-up phase. Approximately 80 patients will be enrolled into this study. Safety evaluations for adverse events, clinical laboratory tests, electrocardiogram and vital signs as well as pharmacokinetic (what the body does to drug) assessments will be conducted in this study. Patients will continue to receive abiraterone acetate plus prednisolone until disease progression or occurrence of unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed adenocarcinoma of the prostate (stage IV)
* Has documented Prostate Specific Antigen (PSA) progression according to protocol-specific prostate specific antigen working group (PSAWG) eligibility criteria
* Has undergone prior chemotherapy for prostate cancer with regimen(s) containing Docetaxel
* Has an ongoing androgen deprivation with serum testosterone less than 50 ng/dL
* Has not received radiotherapy, chemotherapy, or immunotherapy at least 30 days prior to the treatment
* Eastern Cooperative Oncology Group Performance Status less than or equal to 2

Exclusion Criteria:

* Active or uncontrolled autoimmune disease that may require corticosteroid therapy
* Serious or uncontrolled co-existent non-malignant disease, including active and uncontrolled infection
* Uncontrolled hypertension
* Hemoglobin less than or equal to 9.0 g/dL independent of transfusion
* Has abnormal liver function tests
* Surgery or local prostatic intervention within 30 days of the first dose

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2011-08-30 (Actual); Primary Completion 2013-01-24 (Actual); Study Completion 2018-03-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (8):
- South Korea (4):
  - Busan
  - Cheongju-si
  - Seongnam-Si, Gyeonggi-Do
  - Seoul
- Taiwan (4):
  - Kaohsiung City
  - Taichung
  - Taipei
  - Taoyuan

RESULTS

PARTICIPANT FLOW:
Groups:
- Abiraterone Acetate: Abiraterone acetate 1,000 milligram (mg) (administered as 4 * 250 mg tablets) orally once daily at least 1 hour before or 2 hours after a meal, and prednisolone 5 mg orally twice daily until documentation of disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Abiraterone Acetate
Started | 82
Completed | 0
Not Completed | 82
Not completed — Adverse Event | 7
Not completed — Death | 1
Not completed — Withdrawal by Subject | 19
Not completed — Protocol Violation | 2
Not completed — Physician Decision | 13
Not completed — Other | 7
Not completed — Progressive Disease | 32
Not completed — Noncompliance with Study Drug | 1

BASELINE CHARACTERISTICS:
Arm/Group | Abiraterone Acetate
Number analyzed (Participants) | 82
Age, Continuous [Mean (Standard Deviation); unit: years] | 71 (7.35)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 82
Region of Enrollment [Count of Participants; unit: Participants]
  Korea, Republic Of | 52
  Taiwan, Province Of China | 30

OUTCOME MEASURES:

1. Secondary Outcome: Overall Survival
Description: Overall survival is defined as the time interval from the date of the first dose to the date of death due to any reason.
Time Frame: Up to 3 Years
Population: Analysis population included all participants who received at least 1 dose of abiraterone acetate.
Measure: Median (95% Confidence Interval); unit: Days
Groups:
- Abiraterone Acetate and Prednisolone: Abiraterone acetate 1,000 milligram (mg) (administered as 4 * 250 mg tablets) orally once daily at least 1 hour before or 2 hours after a meal, and prednisolone 5 mg orally twice daily until documentation of disease progression or unacceptable toxicity.
Arm/Group | Abiraterone Acetate and Prednisolone
Number analyzed (Participants) | 82
Days | 538 [358.0 to 660.0]

2. Secondary Outcome: Time to PSA Progression
Description: Time to PSA progression was measured as the time interval from the date of the first dose to the date of PSA progression as defined in the protocol-specific PSAWG criteria. For participants who have achieved a greater than or equal to (>=) 50% decrease from the baseline PSA, assessment of time to disease progression is when the PSA has increased 50% above the nadir and at a minimum of 5 nanogram/mililiter (ng/mL). For participants without a PSA decrease of this magnitude or without a decrease, the time for progression is calculated at the time a 25% increase from baseline PSA has been achieved.
Time Frame: Up to 28 Months
Population: Analysis population included all participants who received at least 1 dose of abiraterone acetate.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Abiraterone Acetate and Prednisolone
Number analyzed (Participants) | 82
Days | 141 [112.0 to 170.0]

3. Secondary Outcome: Percentage of Participants With Objective Radiographic Response
Description: Percentage of participants with radiographic objective response is defined as the percentage of participants with complete response (CR) or partial response (PR) as best overall response based on reconciled radiographic disease assessment according to RECIST Version 1.0. The CR is disappearance of all lesions. The PR is at least 30 percent decrease in sum of the longest diameter of target lesions or persistence of one or more non-target lesion(s) or/and maintenance of tumor marker level above the normal limits.
Time Frame: Up to 3 Years
Population: Radiographic response-evaluable population included all participants who received at least 1 dose of abiraterone acetate, and had baseline and at least 1 on treatment tumor assessment.
Measure: Number; unit: Percentage of participants
Arm/Group | Abiraterone Acetate and Prednisolone
Number analyzed (Participants) | 49
Percentage of participants | 6.1

4. Secondary Outcome: Serum Testosterone
Description: Median serum testosterone concentration was reported at baseline and End-of-Treatment visit.
Time Frame: Baseline and End-of-Treatment Visit (up to approximately 3 years)
Population: Analysis population included all participants who received at least 1 dose of abiraterone acetate. "n" signifies those participants who were evaluated for this measure at the specified time point.
Measure: Median (Full Range); unit: nanomole per liter
Arm/Group | Abiraterone Acetate and Prednisolone
Number analyzed (Participants) | 82
nanomole per liter
  Baseline | 1.210 [1.21 to 5.02]
  End-of-Treatment Visit: number analyzed (Participants) | 53
  End-of-Treatment Visit | 1.210 [1.21 to 1.79]

5. Secondary Outcome: Dehydroepiandrosterone Sulfate (DHEA-S)
Description: Median DHEA-S concentration was reported at baseline and End-of-Treatment visit.
Time Frame: Baseline and End-of-Treatment Visit (up to approximately 3 years)
Population: as for outcome 4
Measure: Median (Full Range); unit: micromole per liter
Arm/Group | Abiraterone Acetate and Prednisolone
Number analyzed (Participants) | 82
micromole per liter
  Baseline | 0.725 [0.08 to 6.28]
  End-of-Treatment Visit: number analyzed (Participants) | 10
  End-of-Treatment Visit | 0.080 [0.08 to 0.20]

6. Secondary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly.
Time Frame: Up to 3 Years
Population: Analysis population included all participants who received at least 1 dose of abiraterone acetate.
Measure: Number; unit: Participants
Arm/Group | Abiraterone Acetate and Prednisolone
Number analyzed (Participants) | 82
Participants
  AEs | 81
  SAEs | 40

7. Primary Outcome: Percentage of Participants With Prostate-specific Antigen (PSA) Response
Description: The PSA response was evaluated according to Prostate-Specific Antigen Working Group (PSAWG) criterion, which is, greater than or equal to 50 percent decrease in PSA from Baseline during the study, which would be subsequently confirmed by a measurement that is at least 4 or more weeks after initial documentation of PSA response.
Time Frame: Baseline, Month 4
Population: Analysis population included all participants who received at least 1 dose of abiraterone acetate.
Measure: Number; unit: Percentage of participants
Arm/Group | Abiraterone Acetate and Prednisolone
Number analyzed (Participants) | 82
Percentage of participants | 42.7

ADVERSE EVENTS:
Time Frame: Approximately 3 Years
Arm/Group | Abiraterone Acetate
Serious Adverse Events (participants affected / at risk) | 40/82
Other Adverse Events (participants affected / at risk) | 73/82
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Abiraterone Acetate (N=82)
Anaemia (Blood and lymphatic system disorders) | 3
Microvascular coronary artery disease (Cardiac disorders) | 1
Cataract (Eye disorders) | 1
Abdominal discomfort (Gastrointestinal disorders) | 1
Abdominal distension (Gastrointestinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 2
Ileus (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 3
Asthenia (General disorders) | 3
Chest discomfort (General disorders) | 1
Chills (General disorders) | 1
Septic shock (General disorders) | 1
Fatigue (General disorders) | 1
Generalised oedema (General disorders) | 1
Non-cardiac chest pain (General disorders) | 1
Pyrexia (General disorders) | 2
Appendicitis (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 2
Hepatitis A (Infections and infestations) | 1
Herpes zoster (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Pneumonia cryptococcal (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Septic shock (Infections and infestations) | 1
Urosepsis (Infections and infestations) | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 2
Spinal fracture (Injury, poisoning and procedural complications) | 1
Cachexia (Metabolism and nutrition disorders) | 1
Decreased appetite (Metabolism and nutrition disorders) | 2
Diabetes mellitus (Metabolism and nutrition disorders) | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 3
Chest wall mass (Musculoskeletal and connective tissue disorders) | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Central nervous system lesion (Nervous system disorders) | 1
Encephalopathy (Nervous system disorders) | 1
Lethargy (Nervous system disorders) | 1
Dysuria (Renal and urinary disorders) | 1
Haematuria (Renal and urinary disorders) | 2
Pelvi-ureteric obstruction (Renal and urinary disorders) | 1
Renal failure acute (Renal and urinary disorders) | 1
Urinary retention (Renal and urinary disorders) | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2
Drug rash with eosinophilia and systemic symptoms (Skin and subcutaneous tissue disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Abiraterone Acetate (N=82)
Anaemia (Blood and lymphatic system disorders) | 11
Abdominal discomfort (Gastrointestinal disorders) | 7
Abdominal distension (Gastrointestinal disorders) | 5
Abdominal pain (Gastrointestinal disorders) | 6
Constipation (Gastrointestinal disorders) | 14
Dyspepsia (Gastrointestinal disorders) | 7
Nausea (Gastrointestinal disorders) | 18
Vomiting (Gastrointestinal disorders) | 14
Asthenia (General disorders) | 7
Face oedema (General disorders) | 8
Fatigue (General disorders) | 11
Oedema peripheral (General disorders) | 12
Pyrexia (General disorders) | 6
Nasopharyngitis (Infections and infestations) | 10
Upper respiratory tract infection (Infections and infestations) | 8
Urinary tract infection (Infections and infestations) | 5
Alanine aminotransferase increased (Investigations) | 5
Aspartate aminotransferase increased (Investigations) | 7
Blood alkaline phosphatase increased (Investigations) | 8
Weight decreased (Investigations) | 5
Decreased appetite (Metabolism and nutrition disorders) | 10
Hyperglycaemia (Metabolism and nutrition disorders) | 7
Hypokalaemia (Metabolism and nutrition disorders) | 15
Arthralgia (Musculoskeletal and connective tissue disorders) | 6
Back pain (Musculoskeletal and connective tissue disorders) | 19
Bone pain (Musculoskeletal and connective tissue disorders) | 21
Flank pain (Musculoskeletal and connective tissue disorders) | 5
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 13
Pain in extremity (Musculoskeletal and connective tissue disorders) | 12
Dizziness (Nervous system disorders) | 6
Hypoaesthesia (Nervous system disorders) | 6
Insomnia (Psychiatric disorders) | 10
Haematuria (Renal and urinary disorders) | 5
Nocturia (Renal and urinary disorders) | 5
Proteinuria (Renal and urinary disorders) | 8
Cough (Respiratory, thoracic and mediastinal disorders) | 11
Ecchymosis (Skin and subcutaneous tissue disorders) | 6
Hypertension (Vascular disorders) | 15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested in writing, such publication will be withheld for up to an additional 60 days.